CLINICAL TRIAL: NCT00230165
Title: Studies of Interactions Among Normal and Abnormal Blood Cells, and the Vessel Wall, and Studies of Genetic and Functional Basis of Inherited Platelet, White Blood Cell, Red Blood Cell and Coagulation Disorders
Brief Title: The Genetics and Functional Basis of Inherited Platelet, White Blood Cell, Red Blood Cell, and Blood Clotting Disorders.
Status: Recruiting | Type: Observational
Sponsor: Rockefeller University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: BCO-0417/0726; 5R01HL019278-39 (NIH)
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Glanzmann Thrombasthenia
Keywords: Platelets; Erythrocytes; Leukocytes; Coagulation; Thrombosis
MeSH Terms: conditions — Thrombasthenia; Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal: Normal, healthy volunteers 18 years of age or older of either sex and any ethnic background
- Glanzmann thrombasthenia: Patients with Glanzmann thrombasthenia or their relatives, inherited qualitative and/or quantitative platelet disorders, inherited disorders of white blood cells, inherited disorders of coagulation

SUMMARY:
Blood contains red blood cells, white blood cells, and platelets, as well as a fluid portion termed plasma. We primarily study blood platelets, but sometimes we also analyze the blood of patients with red blood cell disorders (such as sickle cell disease), white blood cell disorders, and disorders of the blood clotting factors found in plasma.

Blood platelets are small cell fragments that help people stop bleeding after blood vessels are damaged. Some individuals have abnormalities in their blood platelets that result in them not functioning properly. One such disorder is Glanzmann thrombasthenia. Most such patients have a bleeding disorder characterized by nosebleeds, gum bleeding, easy bruising (black and blue marks), heavy menstrual periods in women, and excessive bleeding after surgery or trauma. Our laboratory performs advanced tests of platelet function and platelet biochemistry. If we find evidence that a genetic disorder may be responsible, we analyze the genetic material (DNA and RNA) from the volunteer, and when possible, close family members to identify the precise defect.

DETAILED DESCRIPTION:
After volunteers and family members agree to participate, they are seen in the Outpatient Research Center by the Principal Investigator or another physician. A detailed history is obtained, a physical examination is performed, and blood is obtained for further tests. Occasionally patients and family members are requested to return for additional tests. If an abnormality is identified with tests conducted in our research laboratory, we advise the volunteer to have the studies repeated in a laboratory certified to conduct tests on patients.

ELIGIBILITY:
Inclusion Criteria:

A. Normal Healthy Volunteers:

1. Normal healthy volunteers
2. 18 years of age or older
3. Either sex
4. Any ethnic background.

B. Patients with Glanzmann thrombasthenia or their relatives, inherited qualitative and/or quantitative platelet disorders, inherited disorders of white blood cells, inherited disorders of coagulation (including von Willebrand disease):

1. Adults and children
2. Either sex
3. Any ethnic background

Exclusion Criteria:

A. Normal Healthy Volunteers:

1. For studies of platelets that may be affected by anti-platelet therapy, ingestion of aspirin or similar medication in the past week.
2. Having given blood in the last 8 weeks such that the current donation would exceed a total of 250 ml for the 8 week period.
3. Having given blood in the past week such that this donation would result in more than 2 donations in one week.

B. Patients with Glanzmann thrombasthenia or their relatives, inherited qualitative and/or quantitative platelet disorders, inherited disorders of white blood cells, inherited disorders of coagulation (including von Willebrand disease).

1. For studies of platelets that may be affected by antiplatelet therapy, ingestion of aspirin or similar medication in the past week
2. If the patient is known to have a hematocrit ≥25 (assay performed in past 3 months), the same blood drawing criteria as in A, with the addition that for children less than 18 years of age, the maximum amount of blood allowed to be donated in an 8 week period is the lesser of 50 ml or 3 ml/kg.
3. If the patient has a hematocrit <25 or if the hematocrit is unknown, the blood drawing limit is the lesser of 20 ml or 1 ml/kg in any 8 week period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: For normal volunteers, we recruit from laboratory personnel and other volunteers from the NYC area. Patients with platelet disorders, coagulation disorders, or white blood cell disorders, are recruited from among patients referred by other physicians to the P.I. for assessment or via the internet.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2005-09; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Platelet aggregation | minutes
  The initial slope of the increase in light transmission after an agonist is added to a cuvette containing platelet-rich plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Coller, MD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- See also: Link to clinical study description — https://www.rucares.org